CLINICAL TRIAL: NCT03560570
Title: Evaluation of Global Coagulation Balance of 57 Patients With Congenital Disorder of Glycosylation Using the Thrombin Generation Assay
Brief Title: Study of Hemostasis in Patients With Congenital Disorder of Glycosylation
Acronym: CDG-Coag
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: CNIL2126725
Record Dates: First submitted 2018-04-06; First posted 2018-06-18 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-06

CONDITIONS: Congenital Disorders of Glycosylation
Keywords: stroke-like; thrombosis; haemorrhages
MeSH Terms: conditions — Congenital Disorders of Glycosylation; Thrombosis; Hemorrhage | interventions — Bleeding Time

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Plasma sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Event group: CDG with antecedent of stroke-like, thrombosis or haemorrhages
  Interventions: Biological: Coagulation assay; Other: Clinical data collection
- Non event group: CDG without antecedent of stroke-like, thrombosis or haemorrhages
  Interventions: Biological: Coagulation assay; Other: Clinical data collection
- Control: Healthy subject
  Interventions: Biological: Coagulation assay; Other: Clinical data collection

INTERVENTIONS:
Biological: Coagulation assay — Conventional coagulation assays: prothrombin time (PT), activated partial thromboplastin time (aPTT), fibrinogen, factor II, FV, FVII, FX, FVIII, FIX, FXI, FXII, d-dimers, antithrombin, protein C, protein S Thrombin generation assay: in presence or not of soluble thrombomodulin
Other: Clinical data collection — At inclusion, we recorded clinical data about the disease (type and form of congenital disorder of glycosylation, and antecedent of microvascular event: thrombosis, stroke-like or hemorrhages)

SUMMARY:
The purpose of this study is to investigate the coagulation balance in a cohort of congenital disorder of glycosylation (CDG) patients using conventional tests combined with an integrated approach of their coagulation disorders in using TGA in the absence or presence of sTM. Thus, investigators aimed to define if the hemostatic balance in CDG patients, is preserved despite of combined deficiencies in both procoagulant and anticoagulant factors.

DETAILED DESCRIPTION:
In CDG, coagulation abnormalities, affecting both pro and anticoagulant factors, could account for onset of acute microvascular events in these patients. In line with this hypothesis, a previous study reported a correlation between low activity of anticoagulant factors and thrombosis, although stroke-like episodes, the most frequent event, were not analyzed in this study. Moreover, the hemostatic balance is usually investigated by global coagulation tests such as the prothrombin time (PT) and the activated partial thromboplastin (aPTT). However, these tests have serious limitations. First, they explore only 5 % of the whole generated thrombin, enough to clot the plasma. In addition, global tests are insensitive to the coagulation inhibitors, especially the PC system which cannot be mobilized in the absence of thrombomodulin (TM). The thrombin generation assay (TGA), is also a global coagulation assay, but it allows exploration of the whole thrombin formation process from its generation to its inhibition. Moreover, combining different analytical conditions, all the anticoagulant systems could be investigated, including antithrombin in basal conditions and the PC system in the presence of soluble TM (sTM)

ELIGIBILITY:
Inclusion Criteria:

-Clinical diagnosis of Congenital Disorder of Glycosylation (CDG)

Exclusion Criteria:

- no exclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: CDG cohort comes from reference center of rares metabolic diseases of Necker-Enfants malades hospital in Paris
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of haemostatic balance using thrombin generation assay | Up to 1 year
  The assessment of thrombin generation in presence or not of soluble thrombomodulin allows to determine a ratio "R" (without units) calculated as follow : ETP (endogenous thrombin potential) with soluble thrombomodulin (nM/min)/basal ETP (nM/min). This ratio reflects the hypocoagulant or hypercoagulant profile.

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Borgel, PharmaD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker Enfants malades, Paris, France

IPD SHARING:
Plan to Share IPD: No